CLINICAL TRIAL: NCT01963312
Title: A Randomised Clinical Trial to Compare Efficacy and Safety of the Transarterial Supraselective Embolization of the Prostate Compared Versus the Transurethral Resection of the Prostate to Treat the Lower Urinary Tract Symptoms Due to Benign Prostatic Hyperplasia.
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of the Transarterial Supraselective Embolization of the Prostate to Treat the Urinary Symptoms.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Miguel Servet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMSECUR-11; 2011-002108-34 (EudraCT Number)
Record Dates: First submitted 2013-10-11; First posted 2013-10-16 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Transurethral Resection of Prostate; Artery Embolization; Benign Prostatic Hyperplasia; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — Transurethral Resection of Prostate

ARMS (2):
- Transarterial Supraselective Embolization (Experimental): Transarterial supraselective embolization of prostatic arteria with Bead Block 300-500 μm
  Interventions: Procedure: Transarterial Supraselective Embolization of the prostate
- Transurethral Resection (Active Comparator): Surgery to remove part of the prostate gland
  Interventions: Procedure: Transurethral Resection of the prostate

INTERVENTIONS:
Procedure: Transarterial Supraselective Embolization of the prostate
  Arms: Transarterial Supraselective Embolization
Procedure: Transurethral Resection of the prostate
  Arms: Transurethral Resection

SUMMARY:
The purpose of this study is to determine whether the transarterial supraselective embolization (TSE) is a technique as effective as transurethral resection of the prostate (TURP) for the treatment of lower urinary tract symptoms associated with benign prostatic hyperplasia (BPH).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of benign prostatic hyperplasia with moderate or severe obstructive lower urinary tract symptoms
* Refractory to medical treatment for at least 6 months
* Qmax (maximum urinary flow) less than 10 mL/second

Exclusion Criteria:

* Patients not candidates for transurethral resection of the prostate (TURP)
* Advanced atherosclerosis and tortuosity of the iliac arteries
* No visualization of the prostatic artery CT angiography study
* Urethral stenosis, detrusor failure or neurogenic bladder
* Glomerular filtration < 30 mL/min
* Presence of malignant tumor
* History of allergy to iodinated contrast
* Patients with any other medical or social condition, deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2014-03; Primary Completion 2018-04 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Maximum urinary flow (Qmax) | 12 months
  Maximum urinary flow (Qmax) measured prior intervention and one year later

SECONDARY OUTCOMES:
International Prostate Symptom Score (IPSS) measured before and after the intervention | 12 months
Reduction in prostate volume | 12 months
Sexual function | 12 months
  Assessed by International Index of Erectile Function (IIEF) prior and and one year after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Saturnino Napal, MD, Study Director — Complejo Hospitalario de Navarra
Locations (1):
- Complejo Hospitalario de Navarra, Pamplona, Navarre, Spain

REFERENCES:
- [Background] DeMeritt JS, Elmasri FF, Esposito MP, Rosenberg GS. Relief of benign prostatic hyperplasia-related bladder outlet obstruction after transarterial polyvinyl alcohol prostate embolization. J Vasc Interv Radiol. 2000 Jun;11(6):767-70. doi: 10.1016/s1051-0443(07)61638-8. No abstract available. PMID 10877424
- [Background] Carnevale FC, Antunes AA, da Motta Leal Filho JM, de Oliveira Cerri LM, Baroni RH, Marcelino AS, Freire GC, Moreira AM, Srougi M, Cerri GG. Prostatic artery embolization as a primary treatment for benign prostatic hyperplasia: preliminary results in two patients. Cardiovasc Intervent Radiol. 2010 Apr;33(2):355-61. doi: 10.1007/s00270-009-9727-z. Epub 2009 Nov 12. PMID 19908092
- [Background] Pisco J, Campos Pinheiro L, Bilhim T, Duarte M, Rio Tinto H, Fernandes L, Vaz Santos V, Oliveira AG. Prostatic arterial embolization for benign prostatic hyperplasia: short- and intermediate-term results. Radiology. 2013 Feb;266(2):668-77. doi: 10.1148/radiol.12111601. Epub 2012 Nov 30. PMID 23204546
- [Background] Mauro MA. Can hyperplastic prostate follow uterine fibroids and be managed with transcatheter arterial embolization? Radiology. 2008 Mar;246(3):657-8. doi: 10.1148/radiol.2463071721. PMID 18309010
- See also: Related Info — http://www.navarrabiomed.es